CLINICAL TRIAL: NCT00010010
Title: A Phase II Study of the Combination of Exemestane and Goserelin in Premenopausal Women With Metastatic Hormone Receptor Positive Breast Cancer
Brief Title: Exemestane Plus Goserelin in Treating Premenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068431; NYU-0004; P-UPJOHN-NYU-0004; NCI-G00-1906
Record Dates: First submitted 2001-02-02; First posted 2004-04-21 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Goserelin

INTERVENTIONS:
Drug: exemestane
Drug: goserelin acetate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane plus goserelin may fight breast cancer by reducing the production of estrogen.

PURPOSE: Phase II trial to study the effectiveness of exemestane and goserelin in treating premenopausal women who have metastatic breast cancer that has not responded to previous tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of exemestane and goserelin in premenopausal women with hormone receptor positive metastatic breast cancer after tamoxifen failure. II. Determine the toxicity of this regimen in these patients. III. Determine the hormonal profile of patients treated with this regimen. IV. Determine the predictive value of HER-2, epidermal growth factor receptor, and estrogen receptor for response in patients treated with this regimen.

OUTLINE: Patients receive oral exemestane daily on days 1-28 and goserelin subcutaneously on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 22-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic breast cancer that has failed prior tamoxifen therapy Measurable disease No CNS metastases Hormone receptor status: Estrogen or progesterone receptor positive At least 10 fmol/L by biochemical assay OR At least 10% of cells positive by immunochemistry

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Premenopausal defined as estradiol at least 30 pg/mL, follicle stimulating hormone less than 25 mIU/mL, and luteinizing hormone less than 15 mIU/mL Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST no greater than 3 times normal Renal: Stable renal function Pulmonary: No pulmonary embolism Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective non-hormonal contraception during and for 12 weeks after study No other prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix No known hypersensitivity to luteinizing hormone releasing hormone (LHRH), LHRH agonist analogues, or any of the components of goserelin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 2 prior chemotherapy regimens Endocrine therapy: See Disease Characteristics No prior hormonal therapy for metastatic breast cancer No concurrent estrogen (hormone replacement) therapy No other concurrent hormonal agents for breast cancer (e.g., tamoxifen, anastrozole, letrozole, aminoglutethimide, or megestrol) No concurrent corticosteroids for breast cancer unless already receiving such therapy at study entry Radiotherapy: Not specified Surgery: Not specified Other: Concurrent bisphosphonates allowed for bone disease provided measurable disease in non-osseous sites No concurrent anticoagulant therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hamilton, MD, FRACP, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States